CLINICAL TRIAL: NCT04419233
Title: A Multicenter, Non-Interventional, Postmarketing Surveillance Study of Nusinersen Sodium Injection When Used in Routine Medical Practice in China
Brief Title: Non-Interventional, Postmarketing Surveillance Study of Nusinersen Sodium Injection
Acronym: PANDA
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 232SM402
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with 5q SMA and who were prescribed with nusinersen sodium injection in China according to the local marketing authorization.
  Interventions: Drug: Nusinersen Sodium Injection

INTERVENTIONS:
Drug: Nusinersen Sodium Injection — Administered as specified in the treatment arm.
  Other Names: BIIB058; ISIS 396443; Spinraza

SUMMARY:
The primary objective of this study is to evaluate the safety of nusinersen sodium injection in the postmarketing setting in China.The secondary objectives are to collect data on the efficacy and the pharmacokinetics of nusinersen sodium injection in the post-marketing setting in China.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of the participant or his/her legally authorized representative (e.g., parent or legal guardian), as appropriate and applicable, to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations.
* The decision to newly prescribe nusinersen sodium injection according to the local marketing authorization, including documentation of 5q SMA diagnosis, has been made by the Investigator and agreed to by the participant (or legally authorized representative)

Key Exclusion Criteria:

* Hypersensitivity to the active substance or any of the excipients of nusinersen sodium injection.
* Current or past administration of nusinersen sodium injection, in either a commercial or a clinical study setting.
* Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the participant unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are prescribed nusinersen sodium injection in China according to the local marketing authorization (including documentation of 5q SMA diagnosis), agree to the collection and use of data as specified in the protocol, and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 0 up to End of Treatment (2 Years)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event.

SECONDARY OUTCOMES:
Percentage of Participants who Achieved World Health Organization (WHO) Motor Milestone | Baseline, Day 63 and Every 4 Months Up to End of Treatment (2 years)
  WHO Multicentre Growth Reference Study (MGRS), a component to assess gross motor development and is usually assessed in terms of age of achievement of motor milestones. Six distinct gross motor milestones criteria are as follows: sitting without support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone, and walking alone.
Hammersmith Infant Neurological Examination (HINE) Section 2 Scores | Baseline, Day 63 and Every 4 Months Up to End of Treatment (2 years)
  Section 2 of the HINE is used to assess motor milestones of the participants. It is composed of 8 motor milestone categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, and walking.
Number of Participants with Ventilatory Support | Baseline, Day 63 and Every 4 Months Up to End of Treatment (2 years)
Plasma Concentrations of Nusinersen Sodium Injection | Pre-dose and multiple time points post-dose on Day 0, post-dose on Day 28 and pre-dose every 4 months up to end of treatment (2 years)
Cerebrospinal Fluid (CSF) Concentrations of Nusinersen Sodium Injection | pre-dose on Day 0, Day 63, and Every 4 Months Up to End of Treatment (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (9):
- China (9):
  - Research Site, Xicheng, Beijing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Suzhou, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Minhang, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Beijing, Xicheng
  - Research Site, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Jiang Y, Wang Y, Xiong H, Li W, Luo R, Chen W, Yin F, Lu J, Liang J, Chen WJ, Lu X, Wang H, Tang J, Monine M, Makepeace C, Jin X, Foster R, Chin R, Berger Z. A Post-Marketing Surveillance Study of Nusinersen for Spinal Muscular Atrophy in Routine Medical Practice in China: Interim Results. Adv Ther. 2024 Jul;41(7):2743-2756. doi: 10.1007/s12325-024-02852-7. Epub 2024 May 9. PMID 38722537